CLINICAL TRIAL: NCT07358442
Title: A Comparative Clinical Study Assessing Dentin Thickness and Discoloration in Deep Carious Lesions Treated With Biodentine Alone Versus Diode Laser Pre-treatment Followed by Biodentine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Collaborators: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MREC-IRB-03441225
Record Dates: First submitted 2026-01-02; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-07

CONDITIONS: Patients With Deep Carious Lesions; Deep Caries Lesion of Pemanent Teeth; Deep Carious Lesion
Keywords: Vital pulp therapy; Biodentine; Diode laser; Cone beam computed tomography; Dentin bridge; Tooth discoloration; Pulp vitality; Deep carious lesions
MeSH Terms: conditions — Tooth Discoloration | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine Group (Active Comparator): Caries Removal Technique:
  * Caries removal will follow the selective caries removal to soft dentin technique.
  * Occlusal undermined enamel will be eliminated using a #245 high-speed carbide bur to improve visibility and access.
  * A spoon excavator will be used to remove soft, infected dentin from the cavity walls and floor.
  * Firm, discolored, but leathery dentin near the pulp will be removed with a slow-speed sterile carbide round bur to minimize pulp exposure risk.
  * In cases of mechanical pinpoint pulp exposure, minimal bleeding will be controlled using a wet cotton pellet followed by a dry pellet with gentle pressure.
    • Pulp Protection:
  * Biodentine capsule (Septodont, Sain- Maur-des-Fosses, France) will be mixed and placed directly over the exposure site according to the manufacturer's instructions.
  * Application of Biodentine on the exposure site as following ; first keeping the capsule in upright position to remove the white cap and place the open capsule into the stand and ope
  Interventions: Other: Biodentin
- Diode Laser + Biodentine Group (Experimental): * Caries Removal Technique:
    o Identical to Group 1, including selective caries removal and hemostasis measures upon exposure.
  * Diode Laser Application:
    * A 940 nm diode laser (EPIC X™, BIOLASE, USA) will be used immediately after exposure control.
    * Laser Parameters:
      * Wavelength: 940 nm
      * Output Power: 0.1 W
      * Mode: Continuous Wave
      * Duration: 10 seconds
      * Spot Size: 200 µm fiber tip
      * Technique: Non-contact, sweeping motion across the exposure site at a distance of approximately 1 mm from the pulp surface.
    * Safety Measures:
      * All individuals present (patient, operator, assistant) will wear laser-specific protective goggles.
      * Laser warning signs will be displayed to ensure no interruption during application.
      * The laser unit will be calibrated prior to each use, and its output power will be verified using a laser power meter.
  * Pulp Protection:
    * Following laser application, Biodentine will be applied to the exposure site then restored the same as biodentin group
  Interventions: Device: Diode laser

INTERVENTIONS:
Other: Biodentin — Caries removal performed according to standard clinical protocol, followed by direct placement of Biodentine in the cavity. No laser pre-treatment applied.
  Arms: Biodentine Group
Device: Diode laser — Deep carious lesions are treated with diode laser pre-treatment (A 940 nm diode laser (EPIC X™, BIOLASE, USA) will be used immediately after exposure control.
  o Laser Parameters:
  * Wavelength: 940 nm
  * Output Power: 0.1 W
  * Mode: Continuous Wave
  * Duration: 10 seconds
  * Spot Size: 200 µm fiber tip
  * Technique: Non-contact, sweeping motion across the exposure site at a distance of approximately 1 mm from the pulp surface) followed by placement of Biodentine according to standard clinical protocol.
  Arms: Diode Laser + Biodentine Group

SUMMARY:
This interventional clinical study aims to compare dentin thickness preservation and tooth discoloration in deep carious lesions treated with Biodentine alone versus diode laser pre-treatment followed by Biodentine. Participants with deep carious lesions will be allocated to one of two treatment protocols, and clinical and radiographic assessments will be performed to evaluate outcomes. The findings of this study may provide evidence on whether diode laser pre-treatment offers additional clinical benefits when used prior to Biodentine application in the management of deep caries.

DETAILED DESCRIPTION:
Deep carious lesions present a clinical challenge due to the need to remove infected dentin while preserving pulp vitality and preventing postoperative complications. Contemporary minimally invasive dentistry emphasizes selective caries removal and the use of bioactive materials to promote pulp healing and reparative dentin formation.

Biodentine is a calcium silicate-based bioactive cement widely used in vital pulp therapy and indirect pulp capping. It provides favorable sealing ability, biocompatibility, and the potential to stimulate reparative dentinogenesis. However, concerns remain regarding the preservation of dentin thickness and the risk of postoperative tooth discoloration when used in deep cavities.

Diode lasers have been introduced as an adjunctive modality in deep caries management due to their antimicrobial effects, ability to achieve hemostasis, and potential to modify dentin surface characteristics prior to placement of restorative materials. Laser pre-treatment may therefore influence clinical outcomes when used before Biodentine application.

This randomized controlled clinical trial is designed to compare two treatment approaches for deep carious lesions in vital posterior teeth. In the control group, selective caries removal will be performed followed by placement of Biodentine. In the experimental group, diode laser pre-treatment of the cavity will be applied prior to Biodentine placement. All procedures will be carried out under rubber dam isolation and standardized aseptic conditions.

Changes in dentin thickness and radiographic density of the remaining dentin will be evaluated using cone beam computed tomography at baseline and during follow-up visits at 3 and 6 months. Tooth color changes will be assessed using standardized digital photography and spectrophotometric analysis. Pulp vitality will be evaluated using cold testing and electric pulp testing, and periapical clinical status will be assessed through percussion, palpation, and tooth mobility examination.

The primary objective of this study is to compare changes in dentin thickness between Biodentine alone and diode laser pre-treatment followed by Biodentine. Secondary objectives include evaluation of radiographic dentin density, tooth color changes, pulp vitality status, and periapical clinical status over a 6-month follow-up period.

This study aims to determine whether diode laser pre-treatment provides additional clinical benefit when used prior to Biodentine application in the management of deep carious lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged [ 18-45 years] requiring treatment for a single deep carious lesion and willing to provide informed consent and comply with follow-up appointments. Candidates with good general health.
2. tooth-related criteria included reversible pulpitis or asymptomatic restorable vital permanent posterior molar. (based on clinical and radiographic examination, pulp vitality tests).
3. Radiographic evidence of deep caries approaching the pulp (e.g., inner half of dentin).
4. No signs of irreversible pulpitis or periapical pathology.

Exclusion Criteria:

1. Patients undergoing orthodontic treatment or with significant periodontal disease affecting the study tooth or who cannot tolerate CBCT scanning.
2. patients who are medically compromised (systemic diseases affecting bone metabolism or healing (e.g., uncontrolled diabetes)).
3. pregnant ladies, patients with allergy to any component of Biodentine or other materials used, and patients who are not cooperative.
4. Tooth-related criteria involved teeth that have irreversible pulpitis or necrotic pulp (based on symptoms and vitality tests; spontaneous pain, or sustained pain after vitality tests (electrical or cold tests), teeth with pain on percussion ).
5. Teeth with periapical radiolucency and have been already restored before (previous endodontic treatment)
6. Extensive tooth destruction requiring full coronal coverage.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Dentin Thickness | 3 and 6 months
  To evaluate and compare the change in dentin thickness in deep carious lesions treated with Biodentine alone versus diode laser pre-treatment followed by Biodentine using cone beam computed tomography (CBCT).
  Cranex 3D, Soredex, Finland CBCT machine will be used to assess the dentin thickness in Millimeters (mm) by using the linear measurement tool and measuring the distance from the base of restoration to the pulp on sagittal, coronal or cross sectional images generated from CBCT scans after orientation of the orthogonal planes using the software vertical and horizontal reference lines
Radiographic Density of Remaining Dentin | 3 months and 6 months
  To evaluate and compare the radiographic density of the remaining dentin beneath deep carious lesions treated with Biodentine alone versus diode laser pre-treatment followed by Biodentine using CBCT density measurement tools with Gray scale value (CBCT density units).

SECONDARY OUTCOMES:
Change in Tooth Color (ΔE) | 3 and 6 months
  To assess and compare the change in tooth color in teeth treated with Biodentine alone versus diode laser pre-treatment followed by Biodentine using standardized digital photography and spectrophotometric analysis. The total color difference (ΔE) will be calculated based on the CIE L*a*b* color system.
Pulp Vitality Status | 3 and 6 months
  To assess and compare pulp vitality status (vital/ non vital) as binary outcome in both treatment groups using cold stimulus testing and electric pulp testing.
Periapical Clinical Status | 3 months and 6 months
  To assess and compare periapical clinical status as binary outcome (Presence or absence of clinical signs and symptoms) in both groups using percussion, palpation, and tooth mobility examination.

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Center, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared publicly because this is an investigator-initiated academic study conducted at the National Research Centre. Data sharing is restricted by institutional policies and the conditions of ethics committee approval, and the informed consent obtained from participants does not include permission for public sharing of individual-level data.